CLINICAL TRIAL: NCT03018626
Title: Study of R-ACVBP and DA-EPOCH-R in Patients With Newly Diagnosed Non-germinal Center B-cell-like Diffuse Large B-cell Lymphoma
Brief Title: R-ACVBP and DA-EPOCH-R in Patients With Non-GCB DLBCL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Ru Feng, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFL2016-B1
Record Dates: First submitted 2016-11-02; First posted 2017-01-12 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: Non-germinal b-cell-like; R-ACVBP; DA-EPOCH-R
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Etoposide; Doxorubicin; Vincristine; Cyclophosphamide; Prednisone; Vindesine; Bleomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DA-EPOCH-R (Active Comparator): DA-EPOCH-R regimen: rituximab (375 mg/m2) given intravenously (IV) on day 0, etoposide(50 mg/m2), doxorubicin(10 mg/m2) and vincristine(0.4 mg/m2) given continuous intravenously (CIV) from day 1-4(96 hours), cyclophosphamide(750 mg/m2)/dayg IV on days 5, prednisone (60 mg/m2) given orally bid on days 1 through to 5.All patients received granulocyte colony-stimulating factor (G-CSF) beginning on day 6 and continued until the ANC was more than 5 × 109/L above the nadir level. The adjustment paradigm was based on the ANC nadir in the previous cycle as previously described(Wilson, Grossbard et al. 2002)
  Interventions: Drug: Rituximab; Drug: Etoposide; Drug: Doxorubicin; Drug: Vincristine; Drug: Cyclophosphamide; Drug: Prednisone
- Modified R-ACVBP (Experimental): R-ACVBP regimen: rituximab (375 mg/m2) given intravenously (IV) on day 0, doxorubicin (75 mg/m2) and cyclophosphamide (1,200 mg/m2) given intravenously (IV) on day 1, vindesine (2 mg/m2) given on days 1 and 5, bleomycin (10 mg) given IV on days 1 and 5, prednisone (60 mg/m2) given orally on days 1 through to 5.
  Interventions: Drug: Rituximab; Drug: Prednisone; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Vindesine; Drug: Bleomycin

INTERVENTIONS:
Drug: Rituximab — rituximab (375 mg/m2) given intravenously (IV) on day 0
Drug: Etoposide — Etoposide(50 mg/m2) given continuous intravenously (CIV) from day 1-4(96 hours)
  Arms: DA-EPOCH-R
Drug: Doxorubicin — Doxorubicin(10 mg/m2) given continuous intravenously (CIV) from day 1-4(96 hours)
  Arms: DA-EPOCH-R
Drug: Vincristine — Vincristine(0.4 mg/m2) given continuous intravenously (CIV) from day 1-4(96 hours)
  Arms: DA-EPOCH-R
Drug: Cyclophosphamide — Cyclophosphamide(750 mg/m2)/dayg IV on days 5
  Arms: DA-EPOCH-R
Drug: Prednisone — prednisone (100 mg) given orally bid on days 1 through to 5.
Drug: Doxorubicin — Doxorubicin (75 mg/m2) given intravenously (IV) on day 1,
  Arms: Modified R-ACVBP
Drug: Cyclophosphamide — Cyclophosphamide (1,200 mg/m2) given intravenously (IV) on day 1,
  Arms: Modified R-ACVBP
Drug: Vindesine — Vindesine (2 mg/m2) given on days 1 and 5
  Arms: Modified R-ACVBP
Drug: Bleomycin — Bleomycin (10 mg) given IV on days 1 and 5
  Arms: Modified R-ACVBP

SUMMARY:
This is a randomized, open-label, multi-center, phase 3 study evaluating the efficacy of R-ACVBP and DA-EPOCH-R in patients with newly diagnosed non-germinal b-cell-like diffuse large B-cell lymphoma

DETAILED DESCRIPTION:
Diffuse large B-cell lymphoma (DLBCL) is the most common type of non-Hodgkin's lymphoma. According to Hans' algorithms, DLBCL can be identified as 2 subtypes: germinal b-cell-like(GCB) and non-germinal b-cell-like(non-GCB). Approximately 50 to 60% of diffuse large-B cell lymphoma(DLBCL) was non-GCB subtype DLBCL. Although the introduction of rituximab in immunochemotherapy has dramatically improved the outcome of patients with DLBCL, The survival was still poor in non-GCB DLBCL patients treated with R-CHOP.

The LNH03-2B study has shown that R-ACVBP regimen gave a longer PFS (93% vs. 74% at 3 years, p=0.0074) and a longer OS (97% vs. 83% at 3 years, p=0.0067) than R-CHOP in young patients with non-GCB DLBCL. It also showed that R-ACVBP regimen gave a longer PFS (87% vs. 73% at 3 years, p=0.0074) and a longer OS (92% vs. 84% at 3 years, p=0.0067) than R-CHOP in young low-intermediate risk DLBCL patients. The LNH2003-3 study has shown that in high-risk (2/3 IPI factors) DLBCL patients treated with R-ACVBP followed by auto-ASCT results in a 74% PFS and 76% OS. Hematological toxic effects of the intensive regimen were raised but manageable.

The CALGB study showed that in DLBCL patients at least 18 years of age and at least stage II, DA-EPOCH-R regimen is effective in both GCB and non-GCB subtypes, with a 5-years TTP 67%, EFS 58% and OS 68% in non-GCB subtype DLBCL. It is encouraging that PETHEMA Group study showed that in the long-term follow-up of untreated DLBCL patients with poor prognosis, DA-EPOCH-R achieved a 70.8% EFS and 76.4% OS at 10 years in non-GCB subtype DLBCL.

However the efficacy of R-ACVBP compared to DA-EPOCH-R in patients with newly diagnosed non-germinal b-cell-like diffuse large B-cell lymphoma remains unknown. All the above-mentioned results led us to propose a randomized trial comparing R-ACVBP to DA-EPOCH-R in previously untreated patients with non-GCB DLBCL.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically proven CD20+ diffuse large B cell lymphoma (WHO Classification),
* aaIPI>1,
* Age >18 and < 61 years,
* Negative HIV serologies 4 weeks
* Ability to understand and willingness to sign a written informed consent

Exclusion Criteria:

* Any other histological type of lymphoma. Any history of treated or non-treated indolent lymphoma.
* Central nervous system or meningeal involvement by lymphoma.
* Contraindication to any drug contained in the chemotherapy regimens.
* Any serious active disease (according to the investigator's decision).
* Poor renal function (creatinin level>150µmol/l), poor hepatic function (total bilirubin level>30mmol/l, transaminases>2.5 maximum normal level) unless these abnormalities are related to the lymphoma.
* Poor bone marrow reserve as defined by neutrophils <1.5 G/l or platelets <100 G/l, unless related to bone marrow infiltration.
* Treatment with any investigational drug within 30 days before planned first cycle of chemotherapy and during the study.
* Pregnant or lactating women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 402 (Estimated)
Dates: Start 2017-07-27 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 years

SECONDARY OUTCOMES:
Overall survival | 3 years
Complete remission rate | about 13 weeks after initial chemotherapy
  4 cycles after chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Ru Feng, M.D., Principal Investigator — Department of Hematology, Nanfang Hospital, Southern Medical University
Locations (1):
- Ru Feng, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Wilson WH, Grossbard ML, Pittaluga S, Cole D, Pearson D, Drbohlav N, Steinberg SM, Little RF, Janik J, Gutierrez M, Raffeld M, Staudt L, Cheson BD, Longo DL, Harris N, Jaffe ES, Chabner BA, Wittes R, Balis F. Dose-adjusted EPOCH chemotherapy for untreated large B-cell lymphomas: a pharmacodynamic approach with high efficacy. Blood. 2002 Apr 15;99(8):2685-93. doi: 10.1182/blood.v99.8.2685. PMID 11929754
- [Background] Recher C, Coiffier B, Haioun C, Molina TJ, Ferme C, Casasnovas O, Thieblemont C, Bosly A, Laurent G, Morschhauser F, Ghesquieres H, Jardin F, Bologna S, Fruchart C, Corront B, Gabarre J, Bonnet C, Janvier M, Canioni D, Jais JP, Salles G, Tilly H; Groupe d'Etude des Lymphomes de l'Adulte. Intensified chemotherapy with ACVBP plus rituximab versus standard CHOP plus rituximab for the treatment of diffuse large B-cell lymphoma (LNH03-2B): an open-label randomised phase 3 trial. Lancet. 2011 Nov 26;378(9806):1858-67. doi: 10.1016/S0140-6736(11)61040-4. PMID 22118442
- [Background] Fitoussi O, Belhadj K, Mounier N, Parrens M, Tilly H, Salles G, Feugier P, Ferme C, Ysebaert L, Gabarre J, Herbrecht R, Janvier M, Van Den Neste E, Morschhauser F, Casasnovas O, Ghesquieres H, Anglaret B, Brechignac S, Haioun C, Gisselbrecht C. Survival impact of rituximab combined with ACVBP and upfront consolidation autotransplantation in high-risk diffuse large B-cell lymphoma for GELA. Haematologica. 2011 Aug;96(8):1136-43. doi: 10.3324/haematol.2010.038109. Epub 2011 May 5. PMID 21546499
- [Background] Molina TJ, Canioni D, Copie-Bergman C, Recher C, Briere J, Haioun C, Berger F, Ferme C, Copin MC, Casasnovas O, Thieblemont C, Petrella T, Leroy K, Salles G, Fabiani B, Morschauser F, Mounier N, Coiffier B, Jardin F, Gaulard P, Jais JP, Tilly H. Young patients with non-germinal center B-cell-like diffuse large B-cell lymphoma benefit from intensified chemotherapy with ACVBP plus rituximab compared with CHOP plus rituximab: analysis of data from the Groupe d'Etudes des Lymphomes de l'Adulte/lymphoma study association phase III trial LNH 03-2B. J Clin Oncol. 2014 Dec 10;32(35):3996-4003. doi: 10.1200/JCO.2013.54.9493. Epub 2014 Nov 10. PMID 25385729
- [Background] Wilson WH, Jung SH, Porcu P, Hurd D, Johnson J, Martin SE, Czuczman M, Lai R, Said J, Chadburn A, Jones D, Dunleavy K, Canellos G, Zelenetz AD, Cheson BD, Hsi ED; Cancer Leukemia Group B. A Cancer and Leukemia Group B multi-center study of DA-EPOCH-rituximab in untreated diffuse large B-cell lymphoma with analysis of outcome by molecular subtype. Haematologica. 2012 May;97(5):758-65. doi: 10.3324/haematol.2011.056531. Epub 2011 Dec 1. PMID 22133772
- [Background] Wilson WH, Dunleavy K, Pittaluga S, Hegde U, Grant N, Steinberg SM, Raffeld M, Gutierrez M, Chabner BA, Staudt L, Jaffe ES, Janik JE. Phase II study of dose-adjusted EPOCH and rituximab in untreated diffuse large B-cell lymphoma with analysis of germinal center and post-germinal center biomarkers. J Clin Oncol. 2008 Jun 1;26(16):2717-24. doi: 10.1200/JCO.2007.13.1391. Epub 2008 Mar 31. PMID 18378569
- [Background] Purroy N, Bergua J, Gallur L, Prieto J, Lopez LA, Sancho JM, Garcia-Marco JA, Castellvi J, Montes-Moreno S, Batlle A, de Villambrosia SG, Carnicero F, Ferrando-Lamana L, Piris MA, Lopez A. Long-term follow-up of dose-adjusted EPOCH plus rituximab (DA-EPOCH-R) in untreated patients with poor prognosis large B-cell lymphoma. A phase II study conducted by the Spanish PETHEMA Group. Br J Haematol. 2015 Apr;169(2):188-98. doi: 10.1111/bjh.13273. Epub 2014 Dec 18. PMID 25521006
- [Background] Shiozawa E, Yamochi-Onizuka T, Takimoto M, Ota H. The GCB subtype of diffuse large B-cell lymphoma is less frequent in Asian countries. Leuk Res. 2007 Nov;31(11):1579-83. doi: 10.1016/j.leukres.2007.03.017. Epub 2007 Apr 19. PMID 17448534
- [Background] Gutierrez-Garcia G, Cardesa-Salzmann T, Climent F, Gonzalez-Barca E, Mercadal S, Mate JL, Sancho JM, Arenillas L, Serrano S, Escoda L, Martinez S, Valera A, Martinez A, Jares P, Pinyol M, Garcia-Herrera A, Martinez-Trillos A, Gine E, Villamor N, Campo E, Colomo L, Lopez-Guillermo A; Grup per l'Estudi dels Limfomes de Catalunya I Balears (GELCAB). Gene-expression profiling and not immunophenotypic algorithms predicts prognosis in patients with diffuse large B-cell lymphoma treated with immunochemotherapy. Blood. 2011 May 5;117(18):4836-43. doi: 10.1182/blood-2010-12-322362. Epub 2011 Mar 25. PMID 21441466
- [Background] Lenz G, Staudt LM. Aggressive lymphomas. N Engl J Med. 2010 Apr 15;362(15):1417-29. doi: 10.1056/NEJMra0807082. PMID 20393178